CLINICAL TRIAL: NCT00528528
Title: A Phase IIa Randomized, Open-Label Study of Telaprevir (VX-950) Administered Every 12 or Every 8 Hours in Combination With Either Peg-IFN alfa2a (Pegasys) and Ribavirin (Copegus) or Peg-IFN alfa2b (PegIntron) and Ribavirin (Rebetol) in Treatment-Naive Subjects With Chronic Genotype 1 Hepatitis C Infection
Brief Title: An Open-Label Study of Telaprevir Administered Every 12 or 8 Hours in Combination With One of Two Pegylated Interferons and Ribavirin in Treatment-Naive Genotype 1 Chronic Hepatitis C Participants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tibotec BVBA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR013516; VX-950-TIDP24-C208; 2007-001044-44 (EudraCT Number); NCT00614497 (obsolete NCT alias)
Record Dates: First submitted 2007-09-10; First posted 2007-09-12 (Estimated); Results first posted 2013-05-01 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic Hepatitis C; Genotype 1; Telaprevir; Treatment-naïve; VX-950-C208; VX-950-TiDP24-C208
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — telaprevir; peginterferon alfa-2a; peginterferon alfa-2b; Ribavirin; Capsules

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Telaprevir 750 mg with Peg-IFN-alfa-2a/RBV tablet (Experimental): Telaprevir tablets at the dose of 750 milligram (mg) orally administered every 8 hours (hr) for 12 weeks, in combination with standard treatment composed of pegylated interferon (Peg-IFN)-alfa-2a solution for subcutaneous injection at the dose of 180 microgram per week (mcg/week) and ribavirin (RBV) oral tablets at the dose of 1000-1200 mg/day up to 48 weeks.
  Interventions: Drug: Telaprevir; Drug: Peg-IFN-alfa-2a; Drug: Ribavirin (RBV) tablet
- Telaprevir 750 mg with Peg-IFN-alfa-2b/RBV capsule (Experimental): Telaprevir tablets at the dose of 750 mg orally administered every 8 hr for 12 weeks, in combination with standard treatment composed of Peg-IFN-alfa-2b solution for subcutaneous injection at the dose of 1.5 mcg/kilogram/week (mcg/kg/week) and RBV oral capsules at the dose of 800-1200 mg/day up to 48 weeks.
  Interventions: Drug: Telaprevir; Drug: Peg-IFN-alfa-2b; Drug: Ribavirin (RBV) capsule
- Telaprevir 1125 mg with Peg-IFN-alfa-2a/RBV tablet (Experimental): Telaprevir tablets at the dose of 1125 mg orally administered every 12 hr for 12 weeks, in combination with standard treatment composed of Peg-IFN-alfa-2a solution for subcutaneous injection at the dose of 180 mcg/week and RBV oral tablets at the dose of 1000-1200 mg/day up to 48 weeks.
  Interventions: Drug: Telaprevir; Drug: Peg-IFN-alfa-2a; Drug: Ribavirin (RBV) tablet
- Telaprevir 1125 mg with Peg-IFN-alfa-2b/RBV capsule (Experimental): Telaprevir tablets at the dose of 1125 mg orally administered every 12 hr for 12 weeks, in combination with standard treatment composed of Peg-IFN-alfa-2b solution for subcutaneous injection at the dose of 1.5 mcg/kg/week and RBV oral capsules at the dose of 800-1200 mg/day up to 48 weeks.
  Interventions: Drug: Telaprevir; Drug: Peg-IFN-alfa-2b; Drug: Ribavirin (RBV) capsule

INTERVENTIONS:
Drug: Telaprevir — Oval tablets containing 375 mg of telaprevir for oral administration.
Drug: Peg-IFN-alfa-2a — Solution containing Peg-IFN alfa2a for subcutaneous injection in a pre-filled syringe.
  Arms: Telaprevir 1125 mg with Peg-IFN-alfa-2a/RBV tablet; Telaprevir 750 mg with Peg-IFN-alfa-2a/RBV tablet
Drug: Peg-IFN-alfa-2b — Powder containing Peg-IFN-alfa-2b and solvent for solution for subcutaneous injection in a pre-filled pen.
  Arms: Telaprevir 1125 mg with Peg-IFN-alfa-2b/RBV capsule; Telaprevir 750 mg with Peg-IFN-alfa-2b/RBV capsule
Drug: Ribavirin (RBV) tablet — Tablets containing 200 mg RBV for oral administration.
  Arms: Telaprevir 1125 mg with Peg-IFN-alfa-2a/RBV tablet; Telaprevir 750 mg with Peg-IFN-alfa-2a/RBV tablet
Drug: Ribavirin (RBV) capsule — Capsules containing 200 mg RBV for oral administration.
  Arms: Telaprevir 1125 mg with Peg-IFN-alfa-2b/RBV capsule; Telaprevir 750 mg with Peg-IFN-alfa-2b/RBV capsule

SUMMARY:
The purpose of this study is to explore the efficacy, safety, tolerability, pharmacokinetics (the study of the way a drug enters and leaves the blood and tissues over time), and pharmacokinetic-pharmacodynamic relationships of telaprevir administered in two different doses in combination with two standard therapies commercially available for chronic (lasting a long time) genotype 1 Hepatitis (inflammation of the liver) C virus (HCV) infection.

DETAILED DESCRIPTION:
This is a Phase 2a, open-label (all people know the identity of the intervention), multicenter trial (conducted in more than one center) in participants with chronic genotype 1 HCV infection. The trial consists of a Screening phase of approximately 4 weeks, a treatment phase up to 48 weeks depending on participants' individual virologic response, and a follow-up phase of at least 24 weeks. All participants will receive 12 weeks of telaprevir treatment in combination with standard therapy. At Week 12, telaprevir dosing will end and participants will continue on standard therapy only. Participants will be randomly assigned to receive one of the two different dosage regimens of telaprevir (750 milligram [mg] every 8 hours (hr), or 1125 mg every 12 hr) in combination with standard therapy (pegylated interferon [Peg-IFN]-alfa-2a and ribavirin [RBV] or Peg-IFN-alfa-2b and RBV at the standard doses). Efficacy will be evaluated by HCV Ribonucleic Acid (RNA) values, viral response, viral breakthrough, partial response, early viral kinetics and sustained viral response. Pharmacokinetics, Pharmacokinetic-pharmacodynamic relationship will also be evaluated. Safety will be monitored throughout the study duration.

ELIGIBILITY:
Inclusion Criteria:

* Chronic genotype 1 Hepatitis (inflammation of the liver) C infection
* Never been treated for Hepatitis C Viral (HCV) infection
* No clinically significant lab abnormalities
* Amount of HCV Ribonucleic acid (RNA) in the blood more than 10,000 international units/milliliter (IU/mL) at entry
* Liver biopsy or "Fibroscan" test performed during screening or in the past 3 years

Exclusion Criteria:

* Contra-indications for starting anti-HCV therapy
* History or evidence of liver cirrhosis (serious liver disorder in which connective tissue replaces normal liver tissue, and liver failure often occurs) or decompensated liver disease
* Any evidence of significant liver disease in addition to Hepatitis C
* Infected with Human Immunodeficiency Virus (a life-threatening infection which you can get from an infected person's blood or from having sex with an infected person) or Hepatitis B
* Women who are pregnant (carrying an unborn baby), planning to be pregnant or breastfeeding or the partner of a woman who is pregnant or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2007-10; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec-Virco Virology BVBA Clinical Trial, Study Director — Tibotec BVBA
Locations (24):
- Vienna, Austria
- Belgium (4):
  - Brussels
  - Ghent
  - Leuven
  - Liège
- France (7):
  - Angers
  - Clichy
  - Grenoble
  - Lille
  - Nice
  - Paris
  - Vandœuvre-lès-Nancy
- Germany (7):
  - Cologne
  - Düsseldorf
  - Frankfurt
  - Freiburg im Breisgau
  - Hamburg
  - Hanover
  - Tübingen
- Netherlands (2):
  - Leiden
  - Nijmegen
- Spain (3):
  - Barcelona
  - Madrid
  - Valencia

REFERENCES:
- [Derived] Serfaty L, Forns X, Goeser T, Ferenci P, Nevens F, Carosi G, Drenth JP, Lonjon-Domanec I, DeMasi R, Picchio G, Beumont M, Marcellin P. Insulin resistance and response to telaprevir plus peginterferon alpha and ribavirin in treatment-naive patients infected with HCV genotype 1. Gut. 2012 Oct;61(10):1473-80. doi: 10.1136/gutjnl-2011-300749. Epub 2012 Mar 2. PMID 22387529

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 166 participants who were randomly assigned to treatment, only 161 participants received the study treatment.
Period: Overall Study
Arm/Group | Telaprevir 750 mg With Peg-IFN-alfa-2a/RBV Tablet | Telaprevir 750 mg With Peg-IFN-alfa-2b/RBV Capsule | Telaprevir 1125 mg With Peg-IFN-alfa-2a/RBV Tablet | Telaprevir 1125 mg With Peg-IFN-alfa-2b/RBV Capsule
Started | 40 | 42 | 40 | 39
Ongoing at Time of Cut-off | 0 | 0 | 1 | 0
Completed | 37 | 39 | 37 | 36
Not Completed | 3 | 3 | 3 | 3
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1
Not completed — Ineligible to continue the trial | 0 | 0 | 0 | 1
Not completed — Other | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 1 | 1
Not completed — Ongoing participant | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telaprevir 750 mg With Peg-IFN-alfa-2a/RBV Tablet | Telaprevir 750 mg With Peg-IFN-alfa-2b/RBV Capsule | Telaprevir 1125 mg With Peg-IFN-alfa-2a/RBV Tablet | Telaprevir 1125 mg With Peg-IFN-alfa-2b/RBV Capsule | Total
Number analyzed (Participants) | 40 | 42 | 40 | 39 | 161
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 40 | 41 | 40 | 39 | 160
  >=65 years | 0 | 1 | 0 | 0 | 1
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 46.5 [39.5 to 51] | 45.5 [41 to 51] | 40 [34 to 47.5] | 49 [43 to 54] | 46 [37 to 51]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 22 | 19 | 20 | 81
  Male | 20 | 20 | 21 | 19 | 80
Region of Enrollment [Number; unit: Participants]
  Austria | 1 | 1 | 1 | 3 | 6
  Belgium | 6 | 5 | 8 | 4 | 23
  France | 13 | 17 | 12 | 13 | 55
  Germany | 13 | 11 | 11 | 11 | 46
  Italy | 1 | 3 | 2 | 3 | 9
  Netherland | 1 | 1 | 2 | 1 | 5
  Spain | 5 | 4 | 4 | 4 | 17

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Virologic Response at Week 12
Description: Virologic response was either defined as having undetectable Hepatitis C Virus (HCV) ribonucleic acid (RNA) (i.e., no HCV RNA was detected in the participants' plasma samples) or less than 25 international units/milliliter (IU/mL) HCV RNA (i.e., the participants' plasma samples contained traces of HCV RNA at a concentration below the limit of quantification of the viral load assay or no HCV RNA was detected in the samples).
Time Frame: End of treatment (EOT) (up to Week 48)
Population: Full analysis set (FAS) population included all randomly assigned participants who received at least 1 dose of the study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Telaprevir 750 mg With Peg-IFN-alfa-2a/RBV Tablet | Telaprevir 750 mg With Peg-IFN-alfa-2b/RBV Capsule | Telaprevir 1125 mg With Peg-IFN-alfa-2a/RBV Tablet | Telaprevir 1125 mg With Peg-IFN-alfa-2b/RBV Capsule
Number analyzed (Participants) | 40 | 42 | 40 | 39
Percentage of participants | 92.5 | 88.1 | 92.5 | 87.2

2. Secondary Outcome: Time to First Undetectable Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Level
Description: Virologic response was either defined as having undetectable HCV RNA (i.e., no HCV RNA was detected in the participants' plasma samples) or less than 25 IU/mL HCV RNA (i.e., the participants' plasma samples contained traces of HCV RNA at a concentration below the limit of quantification of the viral load assay or no HCV RNA was detected in the samples).
Time Frame: Baseline (Day 1) up to EOT (up to Week 48)
Population: FAS population included all randomly assigned participants who received at least 1 dose of the study medication.
Measure: Median (Full Range); unit: Days
Groups:
- Telaprevir 750 mg With Peg-IFN-alfa-2a/RBV Tablet: Telaprevir tablets at the dose of 750 mg orally administered every 8 hr for 12 weeks, in combination with standard treatment composed of Peg-IFN-alfa-2a solution for subcutaneous injection at the dose of 180 mcg/week and RBV oral tablets at the dose of 1000-1200 mg/day up to 48 weeks.
- Telaprevir 750 mg With Peg-IFN-alfa-2b/RBV Capsule: Telaprevir tablets at the dose of 750 mg orally administered every 8 hr for 12 weeks, in combination with standard treatment composed of Peg-IFN-alfa-2b solution for subcutaneous injection at the dose of 1.5 mcg/kg/week and RBV oral capsules at the dose of 800-1200 mg/day up to 48 weeks.
Arm/Group | Telaprevir 750 mg With Peg-IFN-alfa-2a/RBV Tablet | Telaprevir 750 mg With Peg-IFN-alfa-2b/RBV Capsule | Telaprevir 1125 mg With Peg-IFN-alfa-2a/RBV Tablet | Telaprevir 1125 mg With Peg-IFN-alfa-2b/RBV Capsule
Number analyzed (Participants) | 40 | 42 | 40 | 39
Days | 22 [8 to 99] | 22.5 [8 to 99] | 22 [2 to 99] | 29 [2 to 169]

3. Secondary Outcome: Number of Participants With Viral Breakthrough at End of Treatment (EOT)
Description: Viral breakthrough was defined as a confirmed increase of more than 1 log 10 in HCV RNA level from the lowest level reached or a confirmed value of HCV RNA more than 100 IU/mL in participants whose HCV RNA was previously less than 25 IU/mL.
Time Frame: EOT (up to Week 48)
Population: FAS population included all randomly assigned participants who received at least 1 dose of the study medication.
Measure: Number; unit: Participants
Arm/Group | Telaprevir 750 mg With Peg-IFN-alfa-2a/RBV Tablet | Telaprevir 750 mg With Peg-IFN-alfa-2b/RBV Capsule | Telaprevir 1125 mg With Peg-IFN-alfa-2a/RBV Tablet | Telaprevir 1125 mg With Peg-IFN-alfa-2b/RBV Capsule
Number analyzed (Participants) | 40 | 42 | 40 | 39
Participants | 1 | 6 | 3 | 4

4. Secondary Outcome: Percentage of Participants With Partial Response
Description: Partial response was defined as having at least 2 log drop in HCV RNA from Baseline, but not having undetectable HCV RNA (i.e., no HCV RNA is detected in the participants' plasma samples).
Time Frame: Baseline (Day 1) up to EOT (up to Week 48)
Population: FAS population included all randomly assigned participants who received at least 1 dose of the study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Telaprevir 750 mg With Peg-IFN-alfa-2a/RBV Tablet | Telaprevir 750 mg With Peg-IFN-alfa-2b/RBV Capsule | Telaprevir 1125 mg With Peg-IFN-alfa-2a/RBV Tablet | Telaprevir 1125 mg With Peg-IFN-alfa-2b/RBV Capsule
Number analyzed (Participants) | 40 | 42 | 40 | 39
Percentage of participants | 5 | 0 | 2.5 | 5.1

5. Secondary Outcome: Change From Baseline in Log 10-Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Values at Week 12
Description: Change from baseline in log 10 of Plasma HCV RNA levels were measured using the COBAS TaqMan HCV test (lower limit of quantification 25 IU/mL). The assay used real-time reverse transcription - polymerase chain reaction (RT-PCR) methodology. HCV RNA samples were taken pre-dose of Peg-IFN administration.
Time Frame: Baseline (pre-dose), Week 12
Population: FAS population included all randomly assigned participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Error); unit: log 10 IU/mL
Arm/Group | Telaprevir 750 mg With Peg-IFN-alfa-2a/RBV Tablet | Telaprevir 750 mg With Peg-IFN-alfa-2b/RBV Capsule | Telaprevir 1125 mg With Peg-IFN-alfa-2a/RBV Tablet | Telaprevir 1125 mg With Peg-IFN-alfa-2b/RBV Capsule
Number analyzed (Participants) | 40 | 42 | 40 | 39
log 10 IU/mL
  Baseline | 6.4 (0.09) | 6.5 (0.10) | 6.4 (0.09) | 6.5 (0.11)
  Change from Baseline at Week 12 | -5.2 (0.24) | -5.4 (0.23) | -4.8 (0.36) | -5.1 (0.29)

6. Secondary Outcome: Change From Baseline in Log 10-Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Values at End of Treatment (EOT)
Description: Change from baseline in log 10 of Plasma HCV RNA levels were measured using the COBAS TaqMan HCV test (lower limit of quantification 25 IU/mL). The assay used real-time reverse transcription - polymerase chain reaction (RT-PCR) methodology.
Time Frame: Baseline (pre-dose), EOT (up to Week 48)
Population: FAS population included all randomly assigned participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Error); unit: log 10 IU/mL
Arm/Group | Telaprevir 750 mg With Peg-IFN-alfa-2a/RBV Tablet | Telaprevir 750 mg With Peg-IFN-alfa-2b/RBV Capsule | Telaprevir 1125 mg With Peg-IFN-alfa-2a/RBV Tablet | Telaprevir 1125 mg With Peg-IFN-alfa-2b/RBV Capsule
Number analyzed (Participants) | 40 | 42 | 40 | 39
log 10 IU/mL | -5.5 (0.14) | -5.2 (0.25) | -5.4 (0.22) | -5.3 (0.23)

7. Secondary Outcome: Percentage of Participants With Sustained Viral Response 24 Weeks After End of Treatment (SVR24)
Description: SVR24 was defined as having undetectable HCV RNA (i.e., no HCV RNA is detected in the participants' plasma samples) at EOT and no confirmed detectable HCV RNA levels between EOT and 24 weeks after the last dose of study medication.
Time Frame: EOT (up to Week 48) and up to 24 weeks after EOT
Population: FAS population included all randomly assigned participants who received at least 1 dose of the study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Telaprevir 750 mg With Peg-IFN-alfa-2a/RBV Tablet | Telaprevir 750 mg With Peg-IFN-alfa-2b/RBV Capsule | Telaprevir 1125 mg With Peg-IFN-alfa-2a/RBV Tablet | Telaprevir 1125 mg With Peg-IFN-alfa-2b/RBV Capsule
Number analyzed (Participants) | 40 | 42 | 40 | 39
Percentage of participants | 85.0 | 81.0 | 82.5 | 82.1

ADVERSE EVENTS:
Time Frame: Baseline up to end of telaprevir treatment (Week 12)
Arm/Group | Telaprevir 750 mg With Peg-IFN-alfa-2a/RBV Tablet | Telaprevir 750 mg With Peg-IFN-alfa-2b/RBV Capsule | Telaprevir 1125 mg With Peg-IFN-alfa-2a/RBV Tablet | Telaprevir 1125 mg With Peg-IFN-alfa-2b/RBV Capsule
Serious Adverse Events (participants affected / at risk) | 5/40 | 1/42 | 4/40 | 1/39
Other Adverse Events (participants affected / at risk) | 40/40 | 41/42 | 39/40 | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Telaprevir 750 mg With Peg-IFN-alfa-2a/RBV Tablet (N=40) | Telaprevir 750 mg With Peg-IFN-alfa-2b/RBV Capsule (N=42) | Telaprevir 1125 mg With Peg-IFN-alfa-2a/RBV Tablet (N=40) | Telaprevir 1125 mg With Peg-IFN-alfa-2b/RBV Capsule (N=39)
Anaemia (Blood and lymphatic system disorders) | 4 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0
Hyperthermia (General disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Telaprevir 750 mg With Peg-IFN-alfa-2a/RBV Tablet (N=40) | Telaprevir 750 mg With Peg-IFN-alfa-2b/RBV Capsule (N=42) | Telaprevir 1125 mg With Peg-IFN-alfa-2a/RBV Tablet (N=40) | Telaprevir 1125 mg With Peg-IFN-alfa-2b/RBV Capsule (N=39)
Fatigue (General disorders) | 15 | 15 | 16 | 15
Influenza like illness (General disorders) | 15 | 19 | 11 | 20
Asthenia (General disorders) | 12 | 16 | 8 | 14
Pyrexia (General disorders) | 8 | 14 | 8 | 11
Chills (General disorders) | 3 | 3 | 5 | 4
Injection site erythema (General disorders) | 3 | 6 | 7 | 7
Feeling cold (General disorders) | 2 | 0 | 0 | 1
Injection site reaction (General disorders) | 1 | 2 | 0 | 2
Irritability (General disorders) | 1 | 3 | 1 | 1
Chest discomfort (General disorders) | 0 | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 25 | 15 | 15 | 14
Pruritus (Skin and subcutaneous tissue disorders) | 16 | 22 | 19 | 22
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 9 | 6 | 6
Erythema (Skin and subcutaneous tissue disorders) | 3 | 3 | 1 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 3 | 2 | 9
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 2
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 18 | 14 | 16 | 23
Diarrhoea (Gastrointestinal disorders) | 10 | 9 | 12 | 13
Vomiting (Gastrointestinal disorders) | 7 | 5 | 7 | 12
Abdominal pain upper (Gastrointestinal disorders) | 5 | 5 | 3 | 5
Dry mouth (Gastrointestinal disorders) | 5 | 5 | 6 | 9
Dyspepsia (Gastrointestinal disorders) | 5 | 3 | 3 | 8
Haemorrhoids (Gastrointestinal disorders) | 4 | 5 | 1 | 3
Anal discomfort (Gastrointestinal disorders) | 3 | 3 | 1 | 3
Pruritus ani (Gastrointestinal disorders) | 3 | 8 | 3 | 4
Constipation (Gastrointestinal disorders) | 2 | 1 | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 4 | 0 | 3
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Gastric disorder (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 17 | 14 | 14 | 20
Leukopenia (Blood and lymphatic system disorders) | 6 | 8 | 8 | 9
Lymphopenia (Blood and lymphatic system disorders) | 3 | 6 | 2 | 3
Neutropenia (Blood and lymphatic system disorders) | 2 | 2 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1 | 2 | 1
Headache (Nervous system disorders) | 13 | 18 | 14 | 16
Dizziness (Nervous system disorders) | 4 | 2 | 0 | 6
Disturbance in attention (Nervous system disorders) | 2 | 2 | 1 | 6
Paraesthesia (Nervous system disorders) | 2 | 1 | 0 | 2
Dysgeusia (Nervous system disorders) | 1 | 2 | 6 | 2
Tremor (Nervous system disorders) | 0 | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 8 | 10 | 7 | 9
Depression (Psychiatric disorders) | 6 | 6 | 4 | 6
Sleep disorder (Psychiatric disorders) | 4 | 3 | 4 | 7
Nervousness (Psychiatric disorders) | 3 | 1 | 3 | 4
Anxiety (Psychiatric disorders) | 2 | 3 | 3 | 3
Depressed mood (Psychiatric disorders) | 2 | 2 | 0 | 1
Libido decreased (Psychiatric disorders) | 1 | 1 | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 7 | 9 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 6 | 9 | 7
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 7 | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 2 | 2
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 2
Weight decreased (Investigations) | 4 | 3 | 2 | 2
Blood uric acid increased (Investigations) | 3 | 3 | 1 | 8
Blood phosphorus decreased (Investigations) | 2 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 2 | 3
Platelet count decreased (Investigations) | 1 | 0 | 1 | 2
Blood bilirubin increased (Investigations) | 0 | 0 | 2 | 3
Prothrombin time prolonged (Investigations) | 0 | 0 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 8 | 4 | 6 | 15
Anorexia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 4
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 5 | 9 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 5 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 3
Nasopharyngitis (Infections and infestations) | 3 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 3 | 1 | 0
Dry eye (Eye disorders) | 3 | 0 | 1 | 2
Vision blurred (Eye disorders) | 1 | 1 | 0 | 3
Tachycardia (Cardiac disorders) | 2 | 3 | 3 | 2
Palpitations (Cardiac disorders) | 1 | 2 | 1 | 3
Vertigo (Ear and labyrinth disorders) | 1 | 2 | 1 | 4
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 2
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
As per revised Protocol dated 21 Dec 2007, Investigator may not submit for publication or presentation, the results of trial without prior written consent of Sponsor. The Investigator agrees to allow at least 45 days for Sponsor to review prepublication manuscript prior to submission to Publisher. In accordance with generally recognized principles of scientific collaboration, co-authorship with any company personnel will be discussed and mutually agreed upon before submission to Publisher.